CLINICAL TRIAL: NCT05932823
Title: Airflow and Hip Prosthesis Infections: A Registry Study Comparing Laminar vs. Turbulent Flow in the Danish Hip Arthroplasty Register.
Brief Title: Does the Type of Ventilation Affect the Risk for Infections After Hip Replacements?
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Jacob Moflag Svensson, MD, MD, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: P-2019-796
Record Dates: First submitted 2023-06-17; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Hip Prosthesis Infection
Keywords: Danish microbiology register; periprosthetic joint infection; laminar airflow; turbulent airflow; airflow; total hip arthroplasty; Danish hip arthroplasty register; ventilation system; total hip replacement; hip prosthesis infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laminar Airflow: total hip arthroplasty performed in an operating room using laminar airflow ventilation system
  Interventions: Other: Laminary airflow
- Turbulent Airflow: total hip arthroplasty performed in an operating room using turbulent airflow ventilation system

INTERVENTIONS:
Other: Laminary airflow — A ventilation system that reduces the number of bacteria in the air compared to conventional ventilation.
  Groups: Laminar Airflow

SUMMARY:
Background: During hip replacement surgery, there is a risk that bacteria in the operating room can cause an infection. To try and reduce this risk, some operating rooms use a special system called laminar airflow (LAF), which reduces the number of bacteria in the air. However, it's not clear if LAF is better than the older system, called turbulent airflow (TAF), for preventing infections.

Aim: The aim of this study is to compare the two airflow systems and see if LAF is better at preventing infections after hip replacement surgery.

Methods: Information from a database containing all hip replacement surgeries done in Denmark between 2010 and 2020 is examined. The number of infections that occur in surgeries done with LAF, which reduces the number of bacteria in the air during surgery, is compared to the number of infections that occur in surgeries done with TAF. To make the results more credible, the data from the hip register was combined with data from the bacterial cultures taken during surgery.

Use and relevance: Infections after hip replacement surgery can be very serious and expensive to treat. Hospitals need to choose the best airflow system to help prevent these infections. This study is important because it gives more accurate information about which system is better at preventing infections and can help hospitals make better choices when they are designing or renovating operating rooms.

DETAILED DESCRIPTION:
Rationale and background

Prosthetic joint infection (PJI) is one of the most feared complication after total hip arthroplasty (THA), with increased mortality and morbidity, as well as a significant cost for society. Since the 1960s, in addition to systemic prophylactic antibiotics and antibiotic-laden bone cement, efforts have been made to make the air in the operating rooms (OR) as clean as possible with filtering and replacement of the air .

This has led to the official current PJI incidence of 0.57-0.80 % in the first year after surgery according to the Danish Hip Arthroplasty Register (DHR) and the Swedish Hip Arthroplasty Register (SHAR), even though the true incidence of PJI probably is about 40 % higher, due to under-registration in the registers following revision surgery .

The risk of PJI is potentially affected by contamination in the OR, patient related risk factors and prosthesis factors. The prosthesis factors include type of implant and implant fixation method. Cemented implants have a lower overall revision rate, although the results are not unanimous when it comes to revision due to PJI.

The risk of contamination in the OR is affected by the cleanliness of the air. There are two different types of ventilation systems used to achieve a clean environment in an OR. The first is turbulent airflow (TAF), where the air is continuously replaced with filtered ultra-clean air that trickles down from the ventilation shaft. The second is laminar airflow (LAF) where the ultra-clean air flows in a single direction, with the goal to prevent particles carrying bacteria, that are floating in the air, to land on the patient or sterile equipment.

LAF decreases the bacterial load significantly in the OR, measured in CFUs. However, the number of CFUs has not been found to correlate with the incidence of PJI in real world data, where most studies show no advantage of LAF compared to TAF. Only one major observational study shows that LAF decreases the risk of infection in a subgroup of LAF . All other register studies show no difference between LAF and TAF or a higher risk for PJI with LAF. There are no randomized, controlled trials (RCTs) comparing modern-day ventilation systems when it comes to the PJI incidence in THAs.

There are no randomized, controlled trials (RCTs) comparing modern-day ventilation systems when it comes to the PJI incidence in THAs. However, in 1982, an RCT was conducted by Lidwell et al., comparing different ultraclean air flow systems, including LAF, with standard operating room ventilation at the time. In this study, there was a significant difference in PJI incidence with 2.2 % PJIs in the standard OR group and 1.0 % in the ultraclean group. However, these standard ORs had much higher bacterial contamination, with a median of 164 CFUs/m3 , compared to modern-day TAF ORs, that have a median ranging from 4,5-22 CFU/m3. The ultraclean group had a median of 2-10 CFUs/m3, thus it resembles modern-day TAF ORs, both in bacterial load and PJI rate .

Due to additional costs in building and maintaining LAF systems, a public analysis was conducted in Denmark in 2011 to compare the cost-effectiveness of LAF and TAF. When considering the estimated annual costs, which included operational expenses, depreciation, and interests, LAF ORs were estimated to cost 508,732 DKK per year, whereas TAF ORs were projected to cost 304,530 DKK per year. As a result, there was an annual cost difference of 204,202 DKK (€27,000) per unit, with LAF being 67 % more expensive than TAF. A PJI was estimated to cost the society around 204,000 DKK in the same year .

An issue in the previous studies on PJI in LAF and TAF are that they are epidemiological and rely solely on the PJI diagnosis reported to the different registers. However, diagnosing a PJI is not always evident in a clinical setting. It has been shown that the DHR is lacking both registration of revisions and later confirmed PJI , and a lack of registered PJI revisions has also been observed in the Swedish hip arthroplasty register (SHAR) .

The PJI diagnosis in the DHR can be greatly improved, if combined with the Danish Microbiology Database (MiBa) . When validating the diagnosis PJI in DHR, the sensitivity was found to be only 67 %. When using an algorithm including data from MiBa, sensitivity increased to 90 %, without providing more false positives. A simplified algorithm utilizing MiBa data exhibited no statistically significant difference when compared to the more extensive algorithm employed in the validation study by Gundtoft et al.. This simplified algorithm, which doesn't require access to medical records, will be applied in the criteria for the primary outcome.

Additionally, previous studies show that one positive bacterial sample at a clinically aseptic revision increases the risk of an occult infection, diagnosed later at a re-revision. This will be investigated as well.

Thus, using these new and well validated methods, the investigators aim to estimate the risk of PJI with LAF versus TAF ventilation better than has been done in previous studies.

Data sources

The Danish Civil Registration System (Centrale Person Register, CPR) contains information including vital status and time of emigration on all Danish residents . All Danish residents and citizens are assigned a unique and permanent individual identification number (CPR number) at birth or upon immigration. It enables an unambiguous linkage between different registers and allows an individual follow-up over time .

The Danish National Patient Register (NPR) collects data of all Danish residents contact to a public hospital, including date, performed examinations or surgical procedures and diagnosis, classified by International Classification of Diseases (ICD) . The data includes both outpatient and inpatient contacts and is linked with the patient's CPR number .

The Danish Hip Arthroplasty Register (DHR) collects data including type of OR ventilation from all THAs performed in Denmark, including primary THAs as well as revisions . It is mandatory for all surgeons performing THAs to report to the register, which results in high completeness. The data is previously validated . In the case of a revision, the surgeon reports the indication immediately after surgery . The revisions performed within 90 and 365 days are located in the DHR, which also contains information from the NPR about revisions.

The Danish Microbiology Database (MiBa) automatically collects all microbiology results from all departments of clinical microbiology in Denmark since 2010, which are then stored electronically using the patient's CPR number as patient identifier . The register completeness is previously validated . The data will more specifically be extracted from the Healthcare-Associated Infections Database - HAIBA, a part of MiBa. The Danish National Prescription Register (DNPR) collects detailed information on redeemed prescriptions in Denmark since 1995. It is previously validated and has a high degree of completeness and is frequently used in epidemiological research .

Income Statistics Register - The register contains income data on more than 160 variables including salaries and savings of people with a Danish income and is widely used in research. Each individual is identified with an unambiguous CPR number .

Danish Education Register - The register has a high coverage on education level, both among people born in Denmark and immigrants and is widely used in research. Each individual is identified with an unambiguous CPR number .

Variables

The investigators will look at several variables and adjust for these where needed. The variables obtained from DHR is body mass index (BMI), age, gender, time of surgery, diagnosis, type of prosthesis and fixation method, whether cement is used and if it contains antibiotics, previous operations on the same hip and ASA score. ASA score and BMI are only available from 2017 and onwards in DHR.

From NPR, concomitant diagnoses will be obtained to produce an Elixhauser comorbidity score, and socioeconomic factors, such as income and education will be obtained from the Danish Income Statistics Register and Education Register.

Elaboration of the methods part:

A follow-up time of 90 and 365 days respectively is chosen, since 90 days is the recommended surveillance period in the United States and is traditionally the limit between early and late infections, whereas it is important to have a follow up of a year not to miss up to 20 % of the infections. At 1 year, 80-90 % of the surgically requiring infections that will occur in the lifetime of the hip prosthesis have taken place. After 1 year, the infection rate drastically decreases and is less likely to be due to contamination during surgery.

The definition of PJI is based on the studies by Gundtoft et al. If, where it has been concluded, that the validity of the PJI diagnosis is greatly improved when using these criteria, which are validated specifically for DHR. The original study by Gundtoft et al. used an extensive algorithm to determine if a PJI was present. However, there was no statistically significant difference between the extensive algorithm and a simplified algorithm, that defines a PJI as two or more positive identical bacterial samples.

The investigators definition is in line with international consensus and does not differ greatly from the definition made by the European Bone and Joint Infection Society (EBJIS) , although erythrocyte sedimentation rate, aspiration of joint fluid, white blood cell count in joint fluid and histological examination of intraoperative tissue biopsies are not routinely used in Denmark. Thus, these criteria are not used. Sinus tract communication with the hip joint or an opening to the hip joint is expected to cause the surgeon to register the diagnosis "infection" in DHR upon revision. Data for this analysis will be extracted from DHR and HAIBA. For the revision surgery to be registered in HAIBA, at least three biopsies at the revision surgery are required, hence this is a part of the criteria.

Aseptic loosening is a separate endpoint, since it has been shown that aseptic loosening might in fact turn out to be a PJI and is thus a point of interest.

A sensitivity analysis is made for a) and b), since Milandt et al. have shown that having one positive intraoperative bacterial culture increases the risk of an occult infection, that is later diagnosed upon re-revision. When there was only one unexpected positive culture (unexpected meaning not registered as PJI in DHR), first-time revisions were associated with an increased relative risk of 2.63 for subsequent re-revision specifically for PJI. However, this association was not observed for the patients with two or more unexpected positive cultures, which were much more likely to receive antibiotics and be treated as PJI, after the microbiology results were obtained. This is most likely, because one positive culture has been interpreted as contamination. A sensitivity analysis is made for c), since DHR only have ASA and BMI registered starting in 2017 and thus this cannot be adjusted for prior in the data prior to 2017.

EBJIS have proposed a term called PJI-likely which include 1 positive unexpected positive culture. PJI-likely is based on international consensus; however, the definition relies on analyses that are not commonly performed in routine practice in Denmark, as stated in the description of the primary endpoint. Since it is not possible to use these criteria in Danish register studies, the investigators have instead decided to do sensitivity analyses based on the validation of infections in the DHR by Gundtoft et al. and the findings of Milandt et al..

Statistical analysis:

Descriptive results for continuous variables will be shown as mean(SD)/median(range) depending on the distribution of the variables. Categorical variables will be presented using frequencies and percentages. Persons operated in LAF and TAF ORs are compared using t-tests/Wilcoxon-tests and chi-square tests, respectively. This is supplemented with cumulative incidence plots showing risk of infection (primary outcome) for LAF and TAF, regarding revision due to other causes and death as competing events. The two groups are compared using Grays test. To fulfill the requirements at Statistics Denmark about data on individual persons, a smooth curve is used to make the plot rather than the statistical correct step-function. Information at time 90 and 365 days after the operation will be presented. This type of plot will be used for all endpoints.

For the primary endpoint, two Cox regression analyses will be performed with the time to PJI as outcome. One model will only cover the first 90 days of follow-up, the other will cover all 365 days of follow-up. Censoring is made at time of revision due to other causes than PJI, death, emigration, and end of follow-up (365 days after operation), whichever comes first.

Bilateral THA will be included in the model as two observations with inclusion of a time-dependent variable conditioning on the status of the other hip . A robust sandwich covariance matrix estimate is used to account for the intrapersonal dependence.

The model will include the following potential confounders:

Education, age, comorbidities, gender, previous hip surgery, primary diagnosis, type of cement, type of fixation, year of surgery, income and duration of surgery. ASA and BMI will be adjusted for in sensitivity analysis c). A direct acyclic graph is used when determining the variables needed to adjust for.

The linearity assumption for continuous confounders is checked by including these as cubic splines with 3 to 7 knots and using the model with lowest AIC, as suggested by Harrell .

The proportional hazards assumption for the Cox-regression models is assessed using plots for the cumulative sum of martingale residuals. If the assumption is violated for the exposure (LAF/TAF), the time-axis will be split into smaller parts in which the assumption is fulfilled, and a separate Cox regression is made for each part. If the proportional hazard assumption is violated for confounders, time-dependent covariates is used for these.

Similar Cox-regression models will be used to analyze both secondary endpoints, as well as for the sensitivity analysis of the primary endpoint.

The assumptions of proportional hazards for these endpoints are checked as described for the model for the primary endpoint.

All tests will be two-sided and a p-value of <0.05 will be considered statistically significant. Statistical analysis will be conducted using SAS version 9.4 (SAS Institute Inc.).

Missingness

Thanks to the Danish registers, there is no loss to follow-up for the primary and secondary endpoints, nor for the endpoints of the sensitivity analyses. Information for most of the confounders is based om mandatory registration in DHR, thus a very limited amount of missing data in the confounders is expected (less than 5 % with missing information about one/several confounders). The missingness is not likely to be associated with the exposure, thus the complete case analysis is expected to be valid .

If the missingness is found to be more pronounced, multiple imputation will be used to create a full analysis data set. The imputation will use 100 samples. Multiple imputation will be made using R (The R Foundation). Results from analysis on the full analysis data set as well as for the complete case analysis will be presented.

ELIGIBILITY:
Inclusion Criteria:

* Primary Total hip arthroplasty performed in Denmark between 2010 and 2020

Exclusion Criteria:

* Tumor or metastasis as indication for total hip arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 18 years or older undergoing total hip artroplasty in Denmark between January 1st 2010 - December 31st 2020, expected to be approximately 11.000 per year.
Sampling Method: Probability Sample
Enrollment: 110000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Revisions due to periprosthetic joint infections at 90 days after surgery | t=90 days
  PJI is defined as revision with 2 or more positive biopsies with the same bacteria in MiBa or revision reported to DHR as PJI at t=90 days.
Revisions due to periprosthetic joint infections at 365 days after surgery | t=365 days
  PJI is defined as revision with 2 or more positive biopsies with the same bacteria in MiBa or revision reported to DHR as PJI at t=365 days.

SECONDARY OUTCOMES:
Revisions due to aseptic loosening at 90 days after surgery | t=90 days
  Aseptic loosening is defined as aseptic loosening being reported to DHR as reason for revision at t=90 days.
Revisions due to aseptic loosening at 365 days after surgery | t=365 days
  Aseptic loosening is defined as aseptic loosening being reported to DHR as reason for revision at t=365 days.
Any revision at 90 days after surgery | t=90 days
  Any revision is defined as revision being reported to DHR at t=90 days.
Any revision at 365 days after surgery | t=365 days
  Any revision is defined as revision being reported to DHR at t=365 days.

OTHER OUTCOMES:
Sensitivity analysis: Alternative PJI diagnosis at 90 days | t=90 days
  Primary revision registered as periprosthetic joint infection to DHR or with one or more positive biopsies of a bacterium at at t=90 days.
Sensitivity analysis: Alternative PJI diagnosis at 365 days | t=365 days
  Primary revision registered as periprosthetic joint infection to DHR or with one or more positive biopsies of a bacterium at at t=365 days.
Sensitivity analysis: Viewing of which patients with 1 positive bacterial culture that receive antibiotics at 90 days | t=90
  Primary revision registered to DHR with 1 positive biopsy of a bacterium AND the prescription of a relevant antibiotic at t=90 days.
Sensitivity analysis: Viewing of which patients with 1 positive bacterial culture that receive antibiotics at 365 days | t=365
  Primary revision registered to DHR with 1 positive biopsy of a bacterium AND the prescription of a relevant antibiotic at t=365 days.
PJI in primary surgery between 2017-2020 at 90 days | t=90
  Analysis for the primary endpoint, but for data collected between 2017-2020, allowing for adjustment for BMI and ASA as possible confounders, as these variables are only registered in this period
PJI in primary surgery between 2017-2020 at 365 days | t=365
  Analysis for the primary endpoint, but for data collected between 2017-2020, allowing for adjustment for BMI and ASA as possible confounders, as these variables are only registered in this period

REFERENCES:
- [Background] Akindolire J, Morcos MW, Marsh JD, Howard JL, Lanting BA, Vasarhelyi EM. The economic impact of periprosthetic infection in total hip arthroplasty. Can J Surg. 2020 Jan 29;63(1):E52-E56. doi: 10.1503/cjs.004219. PMID 31995337
- [Background] Gundtoft PH, Pedersen AB, Varnum C, Overgaard S. Increased Mortality After Prosthetic Joint Infection in Primary THA. Clin Orthop Relat Res. 2017 Nov;475(11):2623-2631. doi: 10.1007/s11999-017-5289-6. Epub 2017 Feb 24. PMID 28236084
- [Background] Wildeman P, Rolfson O, Soderquist B, Wretenberg P, Lindgren V. What Are the Long-term Outcomes of Mortality, Quality of Life, and Hip Function after Prosthetic Joint Infection of the Hip? A 10-year Follow-up from Sweden. Clin Orthop Relat Res. 2021 Oct 1;479(10):2203-2213. doi: 10.1097/CORR.0000000000001838. PMID 34061486
- [Background] Hørder M, Bech M, Ejdrup Andersen S. Sundhedsstyrelsen, Dokumentation af Kvalitet og Standardisering Ventilation på operationsstuer København: Sundhedsstyrelsen, Dokumentation af Kvalitet og Standardisering, 2011 [Internet]. 2011 [cited 2023 May 16]. Available from: http://www.sst.dk/mtv
- [Background] Charnley J, Eftekhar N. Postoperative infection in total prosthetic replacement arthroplasty of the hip-joint. With special reference to the bacterial content of the air of the operating room. Br J Surg. 1969 Sep;56(9):641-9. doi: 10.1002/bjs.1800560902. No abstract available. PMID 5808372
- [Background] Gundtoft PH, Pedersen AB, Schonheyder HC, Moller JK, Overgaard S. One-year incidence of prosthetic joint infection in total hip arthroplasty: a cohort study with linkage of the Danish Hip Arthroplasty Register and Danish Microbiology Databases. Osteoarthritis Cartilage. 2017 May;25(5):685-693. doi: 10.1016/j.joca.2016.12.010. Epub 2016 Dec 13. PMID 27986623
- [Background] Lindgren JV, Gordon M, Wretenberg P, Karrholm J, Garellick G. Validation of reoperations due to infection in the Swedish Hip Arthroplasty Register. BMC Musculoskelet Disord. 2014 Nov 19;15:384. doi: 10.1186/1471-2474-15-384. PMID 25410189
- [Background] Charnley J, Eftekhar N. Penetration of gown material by organisms from the surgeon's body. Lancet. 1969 Jan 25;1(7587):172-3. doi: 10.1016/s0140-6736(69)91188-x. No abstract available. PMID 4178415
- [Background] Tanner J, Parkinson H. Double gloving to reduce surgical cross-infection. Cochrane Database Syst Rev. 2002;(3):CD003087. doi: 10.1002/14651858.CD003087. PMID 12137673
- [Background] Rezapoor M, Alvand A, Jacek E, Paziuk T, Maltenfort MG, Parvizi J. Operating Room Traffic Increases Aerosolized Particles and Compromises the Air Quality: A Simulated Study. J Arthroplasty. 2018 Mar;33(3):851-855. doi: 10.1016/j.arth.2017.10.012. Epub 2017 Oct 16. PMID 29174409
- [Background] Bozic KJ, Lau E, Kurtz S, Ong K, Rubash H, Vail TP, Berry DJ. Patient-related risk factors for periprosthetic joint infection and postoperative mortality following total hip arthroplasty in Medicare patients. J Bone Joint Surg Am. 2012 May 2;94(9):794-800. doi: 10.2106/JBJS.K.00072. PMID 22552668
- [Background] Eka A, Chen AF. Patient-related medical risk factors for periprosthetic joint infection of the hip and knee. Ann Transl Med. 2015 Sep;3(16):233. doi: 10.3978/j.issn.2305-5839.2015.09.26. PMID 26539450
- [Background] Makela KT, Matilainen M, Pulkkinen P, Fenstad AM, Havelin L, Engesaeter L, Furnes O, Pedersen AB, Overgaard S, Karrholm J, Malchau H, Garellick G, Ranstam J, Eskelinen A. Failure rate of cemented and uncemented total hip replacements: register study of combined Nordic database of four nations. BMJ. 2014 Jan 13;348:f7592. doi: 10.1136/bmj.f7592. PMID 24418635
- [Background] McMinn DJ, Snell KI, Daniel J, Treacy RB, Pynsent PB, Riley RD. Mortality and implant revision rates of hip arthroplasty in patients with osteoarthritis: registry based cohort study. BMJ. 2012 Jun 14;344:e3319. doi: 10.1136/bmj.e3319. PMID 22700782
- [Background] Kandala NB, Connock M, Pulikottil-Jacob R, Sutcliffe P, Crowther MJ, Grove A, Mistry H, Clarke A. Setting benchmark revision rates for total hip replacement: analysis of registry evidence. BMJ. 2015 Mar 9;350:h756. doi: 10.1136/bmj.h756. PMID 25752749
- [Background] Dale H, Fenstad AM, Hallan G, Havelin LI, Furnes O, Overgaard S, Pedersen AB, Karrholm J, Garellick G, Pulkkinen P, Eskelinen A, Makela K, Engesaeter LB. Increasing risk of prosthetic joint infection after total hip arthroplasty. Acta Orthop. 2012 Oct;83(5):449-58. doi: 10.3109/17453674.2012.733918. PMID 23083433
- [Background] Liu Z, Liu H, Yin H, Rong R, Cao G, Deng Q. Prevention of surgical site infection under different ventilation systems in operating room environment. Front Environ Sci Eng. 2021;15(3):36. doi: 10.1007/s11783-020-1327-9. Epub 2020 Aug 13. PMID 32874704
- [Background] Knudsen RJ, Knudsen SMN, Nymark T, Anstensrud T, Jensen ET, La Mia Malekzadeh MJ, Overgaard S. Laminar airflow decreases microbial air contamination compared with turbulent ventilated operating theatres during live total joint arthroplasty: a nationwide survey. J Hosp Infect. 2021 Jul;113:65-70. doi: 10.1016/j.jhin.2021.04.019. Epub 2021 Apr 29. PMID 33932555
- [Background] Marsault LV, Ravn C, Overgaard A, Frich LH, Olsen M, Anstensrud T, Nielsen J, Overgaard S. Laminar airflow versus turbulent airflow in simulated total hip arthroplasty: measurements of colony-forming units, particles, and energy consumption. J Hosp Infect. 2021 Sep;115:117-123. doi: 10.1016/j.jhin.2021.06.009. Epub 2021 Jun 25. PMID 34182062
- [Background] Ahl T, Dalen N, Jorbeck H, Hoborn J. Air contamination during hip and knee arthroplasties. Horizontal laminar flow randomized vs. conventional ventilation. Acta Orthop Scand. 1995 Feb;66(1):17-20. doi: 10.3109/17453679508994632. PMID 7863761
- [Background] Squeri R, Genovese C, Trimarchi G, Antonuccio GM, Alessi V, Squeri A, La Fauci V. Nine years of microbiological air monitoring in the operating theatres of a university hospital in Southern Italy. Ann Ig. 2019 Mar-Apr;31(2 Supple 1):1-12. doi: 10.7416/ai.2019.2272. PMID 30994159
- [Background] Alsved M, Civilis A, Ekolind P, Tammelin A, Andersson AE, Jakobsson J, Svensson T, Ramstorp M, Sadrizadeh S, Larsson PA, Bohgard M, Santl-Temkiv T, Londahl J. Temperature-controlled airflow ventilation in operating rooms compared with laminar airflow and turbulent mixed airflow. J Hosp Infect. 2018 Feb;98(2):181-190. doi: 10.1016/j.jhin.2017.10.013. Epub 2017 Oct 24. PMID 29074054
- [Background] Langvatn H, Schrama JC, Cao G, Hallan G, Furnes O, Lingaas E, Walenkamp G, Engesaeter LB, Dale H. Operating room ventilation and the risk of revision due to infection after total hip arthroplasty: assessment of validated data in the Norwegian Arthroplasty Register. J Hosp Infect. 2020 Jun;105(2):216-224. doi: 10.1016/j.jhin.2020.04.010. Epub 2020 Apr 11. PMID 32289383
- [Background] Pedersen AB, Svendsson JE, Johnsen SP, Riis A, Overgaard S. Risk factors for revision due to infection after primary total hip arthroplasty. A population-based study of 80,756 primary procedures in the Danish Hip Arthroplasty Registry. Acta Orthop. 2010 Oct;81(5):542-7. doi: 10.3109/17453674.2010.519908. PMID 20860453
- [Background] Hooper GJ, Rothwell AG, Frampton C, Wyatt MC. Does the use of laminar flow and space suits reduce early deep infection after total hip and knee replacement?: the ten-year results of the New Zealand Joint Registry. J Bone Joint Surg Br. 2011 Jan;93(1):85-90. doi: 10.1302/0301-620X.93B1.24862. PMID 21196549
- [Background] Bischoff P, Kubilay NZ, Allegranzi B, Egger M, Gastmeier P. Effect of laminar airflow ventilation on surgical site infections: a systematic review and meta-analysis. Lancet Infect Dis. 2017 May;17(5):553-561. doi: 10.1016/S1473-3099(17)30059-2. Epub 2017 Feb 17. PMID 28216243
- [Background] Wang Q, Xu C, Goswami K, Tan TL, Parvizi J. Association of Laminar Airflow During Primary Total Joint Arthroplasty With Periprosthetic Joint Infection. JAMA Netw Open. 2020 Oct 1;3(10):e2021194. doi: 10.1001/jamanetworkopen.2020.21194. PMID 33064136
- [Background] Brandt C, Hott U, Sohr D, Daschner F, Gastmeier P, Ruden H. Operating room ventilation with laminar airflow shows no protective effect on the surgical site infection rate in orthopedic and abdominal surgery. Ann Surg. 2008 Nov;248(5):695-700. doi: 10.1097/SLA.0b013e31818b757d. PMID 18948793
- [Background] Lidwell OM, Lowbury EJ, Whyte W, Blowers R, Stanley SJ, Lowe D. Effect of ultraclean air in operating rooms on deep sepsis in the joint after total hip or knee replacement: a randomised study. Br Med J (Clin Res Ed). 1982 Jul 3;285(6334):10-4. doi: 10.1136/bmj.285.6334.10. PMID 6805791
- [Background] Gundtoft PH, Overgaard S, Schonheyder HC, Moller JK, Kjaersgaard-Andersen P, Pedersen AB. The "true" incidence of surgically treated deep prosthetic joint infection after 32,896 primary total hip arthroplasties: a prospective cohort study. Acta Orthop. 2015 Jun;86(3):326-34. doi: 10.3109/17453674.2015.1011983. Epub 2015 Jan 30. PMID 25637247
- [Background] Gundtoft PH, Pedersen AB, Schonheyder HC, Overgaard S. Validation of the diagnosis 'prosthetic joint infection' in the Danish Hip Arthroplasty Register. Bone Joint J. 2016 Mar;98-B(3):320-5. doi: 10.1302/0301-620X.98B3.36705. PMID 26920956
- [Background] Milandt NR, Gundtoft PH, Overgaard S. A Single Positive Tissue Culture Increases the Risk of Rerevision of Clinically Aseptic THA: A National Register Study. Clin Orthop Relat Res. 2019 Jun;477(6):1372-1381. doi: 10.1097/CORR.0000000000000609. PMID 31136437
- [Background] Schmidt M, Pedersen L, Sorensen HT. The Danish Civil Registration System as a tool in epidemiology. Eur J Epidemiol. 2014 Aug;29(8):541-9. doi: 10.1007/s10654-014-9930-3. Epub 2014 Jun 26. PMID 24965263
- [Background] Gundtoft PH, Varnum C, Pedersen AB, Overgaard S. The Danish Hip Arthroplasty Register. Clin Epidemiol. 2016 Oct 25;8:509-514. doi: 10.2147/CLEP.S99498. eCollection 2016. PMID 27822092
- [Background] Pedersen A, Johnsen S, Overgaard S, Soballe K, Sorensen HT, Lucht U. Registration in the danish hip arthroplasty registry: completeness of total hip arthroplasties and positive predictive value of registered diagnosis and postoperative complications. Acta Orthop Scand. 2004 Aug;75(4):434-41. doi: 10.1080/00016470410001213-1. PMID 15370588
- [Background] Chaine M, Gubbels S, Voldstedlund M, Kristensen B, Nielsen J, Andersen LP, Ellermann-Eriksen S, Engberg J, Holm A, Olesen B, Schonheyder HC, Ostergaard C, Ethelberg S, Molbak K. Description and validation of a new automated surveillance system for Clostridium difficile in Denmark. Epidemiol Infect. 2017 Sep;145(12):2594-2602. doi: 10.1017/S0950268817001315. Epub 2017 Jul 10. PMID 28689506
- [Background] Pottegard A, Schmidt SAJ, Wallach-Kildemoes H, Sorensen HT, Hallas J, Schmidt M. Data Resource Profile: The Danish National Prescription Registry. Int J Epidemiol. 2017 Jun 1;46(3):798-798f. doi: 10.1093/ije/dyw213. No abstract available. PMID 27789670
- [Background] Baadsgaard M, Quitzau J. Danish registers on personal income and transfer payments. Scand J Public Health. 2011 Jul;39(7 Suppl):103-5. doi: 10.1177/1403494811405098. PMID 21775365
- [Background] Jensen VM, Rasmussen AW. Danish Education Registers. Scand J Public Health. 2011 Jul;39(7 Suppl):91-4. doi: 10.1177/1403494810394715. PMID 21775362
- [Background] Benchimol EI, Smeeth L, Guttmann A, Harron K, Moher D, Petersen I, Sorensen HT, von Elm E, Langan SM; RECORD Working Committee. The REporting of studies Conducted using Observational Routinely-collected health Data (RECORD) statement. PLoS Med. 2015 Oct 6;12(10):e1001885. doi: 10.1371/journal.pmed.1001885. eCollection 2015 Oct. PMID 26440803
- [Background] Muscatelli S, Zheng H, Muralidharan A, Tollemar V, Hallstrom BR. Limiting the Surveillance Period to 90 Days Misses a Large Portion of Infections in the First Year After Total Hip and Knee Arthroplasty. Arthroplast Today. 2022 May 30;16:90-95. doi: 10.1016/j.artd.2022.04.009. eCollection 2022 Aug. PMID 35662991
- [Background] Tande AJ, Patel R. Prosthetic joint infection. Clin Microbiol Rev. 2014 Apr;27(2):302-45. doi: 10.1128/CMR.00111-13. PMID 24696437
- [Background] Parvizi J, Gehrke T, Chen AF. Proceedings of the International Consensus on Periprosthetic Joint Infection. Bone Joint J. 2013 Nov;95-B(11):1450-2. doi: 10.1302/0301-620X.95B11.33135. PMID 24151261
- [Background] McNally M, Sousa R, Wouthuyzen-Bakker M, Chen AF, Soriano A, Vogely HC, Clauss M, Higuera CA, Trebse R. Infographic: The EBJIS definition of periprosthetic joint infection. Bone Joint J. 2021 Jan;103-B(1):16-17. doi: 10.1302/0301-620X.103B1.BJJ-2020-2417. No abstract available. PMID 33380197
- [Background] Hipfl C, Mooij W, Perka C, Hardt S, Wassilew GI. Unexpected low-grade infections in revision hip arthroplasty for aseptic loosening : a single-institution experience of 274 hips. Bone Joint J. 2021 Jun;103-B(6):1070-1077. doi: 10.1302/0301-620X.103B6.BJJ-2020-2002.R1. PMID 34058865
- [Background] Goldman AH, Osmon DR, Hanssen AD, Pagnano MW, Berry DJ, Abdel MP. The Lawrence D. Dorr Surgical Techniques & Technologies Award: Aseptic Reoperations Within One Year of Primary Total Hip Arthroplasty Markedly Increase the Risk of Later Periprosthetic Joint Infection. J Arthroplasty. 2020 Jun;35(6S):S10-S14. doi: 10.1016/j.arth.2020.02.054. Epub 2020 Feb 28. PMID 32192836
- [Background] Lie SA, Engesaeter LB, Havelin LI, Gjessing HK, Vollset SE. Dependency issues in survival analyses of 55,782 primary hip replacements from 47,355 patients. Stat Med. 2004 Oct 30;23(20):3227-40. doi: 10.1002/sim.1905. PMID 15449328
- [Background] Harrell FE. Regression Modeling Strategies: With Applications to Linear Models, Logistic Regression, and Survival Analysis [Internet]. New York, NY: Springer New York; 2001 [cited 2023 Jun 16]. (Springer Series in Statistics). Available from: http://link.springer.com/10.1007/978-1-4757-3462-1
- [Background] Jakobsen JC, Gluud C, Wetterslev J, Winkel P. When and how should multiple imputation be used for handling missing data in randomised clinical trials - a practical guide with flowcharts. BMC Med Res Methodol. 2017 Dec 6;17(1):162. doi: 10.1186/s12874-017-0442-1. PMID 29207961
- [Background] Lindgren V, Gordon M, Wretenberg P, Karrholm J, Garellick G. Deep infection after total hip replacement: a method for national incidence surveillance. Infect Control Hosp Epidemiol. 2014 Dec;35(12):1491-6. doi: 10.1086/678600. Epub 2014 Oct 24. PMID 25419771
- See also: Danmarks statistik befolkningstal [Internet]. 2022. — https://www.dst.dk/da/Statistik/emner/borgere/befolkning/befolkningstal
- See also: WHO International Classification of Diseases. 2022 Jul 9 — https://www.who.int/classifications/classification-of-diseases
- See also: The Danish Hip Arthroplasty Register (DHR), 2021 National Annual Report. — http://www.dhr.dk
- See also: Statens Serum Institut. Hoftealloplastikinfektion [Internet]. 2023 [cited 2023 May 31]. — https://miba.ssi.dk/overvaagningssystemer/haiba/casedefinitioner/hoftealloplastik

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT05932823/Prot_SAP_000.pdf